CLINICAL TRIAL: NCT02296437
Title: Pilot Study of Transcranial Direct Current Stimulation (tDCS) and Cognitive Task in Depression.
Brief Title: Transcranial Direct Current Stimulation (tDCS) and Cognitive Task in Depression
Acronym: tDCS + CT
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The University of New South Wales (Other)
Collaborators: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Principal Investigator, Melissa Pigot, Research assistant, The University of New South Wales
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HC14216
Record Dates: First submitted 2014-11-18; First posted 2014-11-20 (Estimated); Last update posted 2017-10-17 (Actual); Status verified 2017-10

CONDITIONS: Depression
MeSH Terms: conditions — Depression | interventions — Cognitive Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- tDCS + CT (Experimental)
  Interventions: Other: Transcranial direct current stimulation combined with cognitive training

INTERVENTIONS:
Other: Transcranial direct current stimulation combined with cognitive training

SUMMARY:
Among antidepressant treatments, electroconvulsive therapy (ECT) remains the most effective. However, patient concerns with cognitive side effects have encouraged trials of new, non-convulsive forms of mild brain stimulation such as transcranial Direct Current Stimulation (tDCS). Our past and present studies of tDCS suggest that it has antidepressant effects and is safe, painless and well tolerated. However, not all patients may have an adequate response, raising the need to find ways of optimising efficacy. This clinical pilot study will examine the feasibility and safety of combining tDCS with a cognitive training task which engages the same brain region targeted by tDCS for treatment of depression.

ELIGIBILITY:
Inclusion Criteria:

1. Participants are aged 18-65 years.
2. Participant meets criteria for a DSM-V Major Depressive episode. Criteria are as follows: Five or more symptoms present during the same 2-week period, including either 1 or 2: 1) depressed mood, 2) loss of interest or pleasure, 3) significant weight loss or gain, 4) insomnia or hypersomnia, 5) psychomotor agitation or retardation, 6) fatigue or loss of energy, 7) feelings of worthlessness or excessive or inappropriate guilt, 8) diminished ability to think concentrate or make decisions, and 9) recurrent thoughts of death, recurrent suicidal ideation, suicide attempt or plan.
3. MADRS score of 20 or more.
4. Right handed
5. A history of non-response to ≥ 2 adequate trials of antidepressant medication treatment.

Exclusion Criteria:

1. DSM-V psychotic disorder.
2. Drug or alcohol abuse or dependence (preceding 6 months).
3. Inadequate response to ECT (current episode of depression).
4. Regular benzodiazepine medication
5. Rapid clinical response required, e.g., due to high suicide risk.
6. Clinically defined neurological disorder or insult.
7. Metal in the cranium, skull defects, or skin lesions on scalp (cuts, abrasions, rash) at proposed electrode sites.
8. Pregnancy.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2014-11; Primary Completion 2019-11 (Estimated)

PRIMARY OUTCOMES:
Montgomery and Asberg Depression Rating Scale (MADRS) | 6 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- University of New South Wales, Sydney, New South Wales, Australia